CLINICAL TRIAL: NCT03883516
Title: Improving Emergency Management of Status Epilepticus - a High-fidelity Simulator-based Randomized Controlled Trial
Brief Title: Improving Emergency Management of Status Epilepticus
Acronym: SESIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Requ_2019-00168; me19Sutter3
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Status Epilepticus
Keywords: guideline for the treatment of Status Epilepticus; antiseizure drugs (ASDs)
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No pre-briefing prior to the simulation training (Placebo Comparator): No pre-briefing prior to the simulation training
  Interventions: Other: No Pre-briefing
- Pre-briefing with the current SE treatment guidelines (Active Comparator): pre-briefing with the current SE treatment Guidelines published by the American Epilepsy Society
  Interventions: Other: Pre-briefing with the current SE treatment guidelines
- pre- briefing with consolidated SE treatment guideline (Active Comparator): pre-briefing with the consolidated "one page" SE treatment guideline
  Interventions: Other: Pre-briefing with a consolidated "one page" SE treatment guide

INTERVENTIONS:
Other: Pre-briefing with the current SE treatment guidelines — instruction of the study participants according to the evidence-based guideline for the treatment of SE published by the American Epilepsy Society prior to the simulation training
  Arms: Pre-briefing with the current SE treatment guidelines
Other: Pre-briefing with a consolidated "one page" SE treatment guide — instruction of the study participants with a consolidated "one page" SE treatment guide prior to the simulation training
  Arms: pre- briefing with consolidated SE treatment guideline
Other: No Pre-briefing — no instruction of the study participants prior to the simulation training
  Arms: No pre-briefing prior to the simulation training

SUMMARY:
In the trial the effectiveness of pre-briefing physicians with the current guideline on Status epilepticus (SE) treatment or a consolidated "one page" guideline regarding quality enhancement of the physician's clinical performances is investigated.

DETAILED DESCRIPTION:
Status epilepticus (SE) is a life-threatening neurological emergency defined as a state of continuous seizure or multiple seizures without full recovery of sensory, motor and/or cognitive function for at least 30 minutes. To achieve high quality management of SE, the American Epilepsy Society published an evidence-based guideline for the treatment of SE, which serves as reference for most national guidelines, but analyses regarding practicability, strict adherence, correct translation into clinical practice, and identification of recommended treatment steps at risk of being modified or missed are lacking. Simulator-based studies offer a platform for the design of standardized clinical scenarios that enable detailed investigations regarding the effect of the implementation and practicability of treatment guidelines.

This randomized controlled intervention study performed at the simulation center of the medical intensive care units (ICUs) at the University Hospital Basel is to investigate the effectiveness of pre-briefing physicians with both the current guideline on Status epilepticus (SE) treatment or a consolidated "one page" guideline regarding quality enhancement of the physicians' clinical performances..

Physicians from different medical specialties and with different duration of clinical experience will be enrolled. Participants will be randomly assigned to one of the following three pre-briefing groups: (1) no pre-briefing prior to the simulation training; (2) pre-briefing with the current SE treatment guidelines; (3) pre-briefing with the consolidated "one page" SE treatment guideline.

ELIGIBILITY:
Inclusion Criteria:

* Physicians from different medical specialties working at the University Hospital Basel

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Time to SE recognition (minutes) | from start of simulation training until recognition of seizure and/or SE (max. 20 minutes)
  time to recognition of seizure and/or SE

SECONDARY OUTCOMES:
administration of anti-seizure medication | within the first 20 minutes after beginning of the simulation training
  time of administration of anti-seizure medication (minutes)
dose of anti-seizure medication | within the first 20 minutes after beginning of the simulation training
  dose of anti-seizure medication (mg)
time to correct airways protection | from start of simulation training until correct airways protection (max. 20 minutes)
  time to correct airways protection (minutes)
quantification of Glasgow Coma Score (GCS) | within the first 20 minutes after beginning of the simulation training
  GCS is a neurological scale recording the state of a person's consciousness ; The scale is composed of three tests: eye, verbal and motor responses. The three values separately as well as their sum are considered. The lowest possible GCS (graded 1 in each element) is 3 (deep coma or death), while the highest is 15 (fully awake person).

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. MD, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland